CLINICAL TRIAL: NCT05120362
Title: An Investigator-initiated Trial to Evaluate the Efficacy and Safety of JAK Inhibitor Cream for the Treatment of EGFR-inhibitor-induced Skin Rash
Brief Title: A Study to Evaluate JAK Inhibitor Cream in EGFR-inhibitor-induced Skin Rash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEH002
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Acneiform Eruptions
Keywords: EGFR; Acneiform Rash
MeSH Terms: conditions — Acneiform Eruptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cream containing JAK Inhibitor (Experimental)
  Interventions: Drug: Cream containing JAK Inhibitor

INTERVENTIONS:
Drug: Cream containing JAK Inhibitor — The study drug is a cream containing JAK Inhibitor.

SUMMARY:
Epidermal growth factor receptor inhibitors (EGFRIs) are widely used targeted agents that have been approved for the treatment of various tumor types. In some clinical studies with EGFRIs, the incidence of dermatology AE, the skin rash, is reportedly as high as 95%, which profoundly impact the patients' quality of life. However no treament for onset skin rash has been approved to be effective by any clinical trial yet. Janus kinase (JAK) inhibitor, has been approved for or studied in a variety of skin conditions such as alopecia areata, atopic dermatitis, and psoriasis. Thus the investigators intend to evaluate the efficacy and safety of JAK inhibitor cream for the treatment of EGFRIs-induced skin rash in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Pathologically conﬁrmed cancer receiving EGFRI-based therapy (monotherapy or as part of a combination therapy regimen).
* Skin rash causally related to EGFRI therapy of grade 1 or higher (according to MESTT criteria).
* ECOG performance score < 2.
* Able to use topical medications and complete questionnaires reliably with or without assistance.
* Life expectancy of greater than 6 months.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Use of any other topical medications in the treatment areas (face) within 7 days prior to randomization or duing the study.
* Use of Tetracycline (e.g. minocycline, doxycycline) within 14 days prior to randomization or duing the study.
* Use of other cancer medications known to result in skin rash in the face or upper chest/upper back area within 4 weeks prior to randomization or duing the study.
* Known hypersentitivity to JAK inhibitors.
* With other skin disorders that may affect efficacy evaluation, including but not limited to: eczema, psoriasis, etc.
* Uncontrolled intercurrent illness.
* Significantly abnormal lab test.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of grade 0 or 1 patients at Week 4 | 4 weeks
  Determine the proportion of patients receiving JAK Inhibitor Cream who have achieved 1 or 2 grade(s) decrease in skin rash (according to MASCC EGFR Inhibitor Skin Toxicity Tool - the MESTT criteria for Papulopustular Eruption, which includes 4 grades, Grade 3 as the most severe condition and Grade 0 as no symptom) at Week 4

SECONDARY OUTCOMES:
Proportion of grade 0 or 1 patients at Week 2 | 2 weeks
  Determine the proportion of patients receiving JAK Inhibitor Cream who have achieved 1 or 2 grade(s) decrease in skin rash (according to MASCC EGFR Inhibitor Skin Toxicity Tool - the MESTT criteria for Papulopustular Eruption, which includes 4 grades, Grade 3 as the most severe condition and Grade 0 as no symptom) at Week 2
Proportion of grade 0 or 1 patients at Week 6 | 6 weeks
  Determine the proportion of patients receiving JAK Inhibitor Cream who have achieved 1 or 2 grade(s) decrease in skin rash (according to MASCC EGFR Inhibitor Skin Toxicity Tool - the MESTT criteria for Papulopustular Eruption, which includes 4 grades, Grade 3 as the most severe condition and Grade 0 as no symptom) at Week 6
Change of PRO (FACT-EGFR 14) from baseline at Week 4 | 4 weeks
  Determine the Change of PRO (according to FACT-EGFR 14 Questionnaire, which includes 14 QoL questions & each scoring from 0 to 4, 4 as the most severe condition and 0 as no symptom) from baseline in patients receiving JAK Inhibitor Cream at Week 4
Safety of study drug | 6 weeks
  Safety of study drug as determined by the number of participants with abnormal laboratory values and/or Adverse Events that are related to study treatment, especially local irritation

CONTACTS AND LOCATIONS:
Overall Officials: Nan Xu, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] You Q, Chen L, Li S, Liu M, Tian M, Cheng Y, Xia L, Li W, Yao Y, Li Y, Zhou Y, Ma Y, Lv D, Zhao L, Wang H, Wu Z, Hu J, Ju J, Jia C, Xu N, Luo J, Zhang S. Topical JAK inhibition ameliorates EGFR inhibitor-induced rash in rodents and humans. Sci Transl Med. 2024 Jun 19;16(752):eabq7074. doi: 10.1126/scitranslmed.abq7074. Epub 2024 Jun 19. PMID 38896602